CLINICAL TRIAL: NCT01590238
Title: Enhancing Hair Density With Platelet Rich Fibrin Matrix (PRFM)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: The New York Eye & Ear Infirmary (Other)
Responsible Party: Principal Investigator, Anthony P. Sclafani, Director of Facial Plastic Surgery, The New York Eye & Ear Infirmary
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2012-1
Record Dates: First submitted 2012-04-29; First posted 2012-05-02 (Estimated); Results first posted 2016-11-10 (Estimated); Last update posted 2017-02-15 (Actual); Status verified 2016-12

CONDITIONS: Alopecia
Keywords: alopecia
MeSH Terms: conditions — Alopecia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment with PRFM (Experimental): Subjects treated monthly 3 times with intradermal injections of PRFM into bald/balding scalp. Post-treatment hair density index measured and compared to hair density index measured prior to treatment for each subject.
  Interventions: Biological: PRFM treatment

INTERVENTIONS:
Biological: PRFM treatment — Study participants are treated in the initial visit, and at the 1 and 2 month follow-up visit. 4-8 cc of autologous platelet rich fibrin matrix (PRFM) is isolated from 9-18 cc of peripheral blood. PRFM is then injected intradermally in 0.10 cc aliquots in areas of alopecia for each treatment.

SUMMARY:
Clinical alopecia occurs due to miniaturization of the hair shafts as well as loss of active production of hair shafts. PRFM has been shown to induce dermal angiogenesis, and anecdotal findings of improvement of hair appearance after PRFM injection in the scalp suggest that PRFM may play a role in the treatment of thinning hair. Patients will be treated on a monthly basis with intradermal injections of autologous PRFM for 3 months. Changes in hair density will be assessed by comparing pre- and post-treatment photographs and non-invasive measurements of hair density at 1, 2, 3, 4 and 6 months after initial treatment.

ELIGIBILITY:
Inclusion Criteria:

* age 18- 75 years old
* frontal and/or crown alopecia

Exclusion Criteria:

* bleeding disorder

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2012-05; Primary Completion 2013-09 (Actual); Study Completion 2013-11 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- The New York Eye & Ear Infirmary, New York, New York, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treatment With PRFM
Started | 15
Completed | 13
Not Completed | 2

BASELINE CHARACTERISTICS:
Groups:
- Treatment With PRFM: Subjects with androgenetic alopecia clinically diagnosed were treated monthly 3 times with intradermal injections of PRFM into bald/balding scalp. Post-treatment hair density index measured and compared to hair density index measured prior to treatment for each subject.
  PRFM treatment: Study participants are treated in the initial visit, and at the 1 and 2 month follow-up visit. 4-8 cc of autologous platelet rich fibrin matrix (PRFM) is isolated from 9-18 cc of peripheral blood. PRFM is then injected intradermally in 0.10 cc aliquots in areas of alopecia for each treatment.
Arm/Group | Treatment With PRFM
Number analyzed (Participants) | 15
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.2 (18.2)
Gender [Count of Participants; unit: Participants]
  Female | 6
  Male | 9
Region of Enrollment [Number; unit: participants]
  United States | 15
Hair density index measured prior to intervention [Mean (Standard Deviation); unit: percent of pre treatment value] — Hair density as measured with proprietary hair densitometer in a 2cm x 2cm square in the midline at a predetermined distance from the nasal root (individual measurement but held constant for multiple measurements in the same subject over time).
  percent of pre treatment value | 100 (0)

OUTCOME MEASURES:

1. Primary Outcome: Hair Density Change After Three Treatments
Description: Hair density index at calibrated distance from glabella in a 2 cm x 2 cm midline square at 6 month follow up visit as a percentage of initial (pre-treatment) hair density index, measured using a proprietary hair densitometer.
Time Frame: 6 months after initial visit
Measure: Mean (Standard Deviation); unit: percentage of pre-treatment hair density
Groups:
- Treatment With PRFM: Subjects with androgenetic alopecia clinically diagnosed were treated monthly 3 times with intradermal injections of PRFM into bald/balding scalp. Post-treatment hair density index measured (6 months after initial treatment) and compared to hair density index measured prior to treatment for each subject.
Arm/Group | Treatment With PRFM
Number analyzed (Participants) | 13
percentage of pre-treatment hair density | 175.1 (46.8)

ADVERSE EVENTS:
Time Frame: First six months after initial treatment.
Arm/Group | Treatment With PRFM
Serious Adverse Events (participants affected / at risk) | 0/15
Other Adverse Events (participants affected / at risk) | 0/15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No